CLINICAL TRIAL: NCT07284355
Title: Knowledge, Attitude, Practices and Barriersof General Practitioner RegardingHelicobacter Pylori Diagnosis andTreatment
Brief Title: Barriers of General Practitioner Regarding Helicobacter Pylori.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohanad Abd_Elaleem Sayed Amer, Resident at tropical department., Assiut University
Other Study IDs: Helicobacter pylori
Record Dates: First submitted 2025-09-29; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-09

CONDITIONS: H.Pylori Infection
Keywords: H.pylori infection

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Demographic , knowledge , Practices , attitude and barriers: Section A: demographic data (age, gender, years of experience, workplace) Section B: knowledge (transmission, symptoms, diagnostic methods,. treatment guidelines) Section C: attitude (perceived importance, confidence in diagnosis/treatment) Section D: practice (frequency of testing, treatment regimen used). Section E: barriers (e.g., Lack of resources, guidelines, time constraints, patient adherence)

SUMMARY:
This study aims to evaluate the knowledge, attitudes, and clinical practices of general practitioners regarding the diagnosis and treatment of Helicobacter pylori infection. The study also seeks to identify the main barriers that prevent proper management of the condition. The central hypothesis is that gaps in knowledge and challenges in clinical practice contribute to variations in how general practitioners diagnose and treat H. pylori infection.

DETAILED DESCRIPTION:
This study explores the knowledge, attitudes, and practices of general practitioners regarding the diagnosis and treatment of Helicobacter pylori infection. It also examines the barriers that may affect appropriate clinical decision-making in managing this common gastrointestinal condition. By assessing physicians' understanding of recommended diagnostic techniques, treatment regimens, and follow-up strategies, the study aims to identify areas where education or system-level improvements may be needed.

The study hypothesizes that insufficient knowledge of current guidelines, limited access to diagnostic tests, and patient-related or system-related barriers contribute to inconsistent management of H. pylori infection among general practitioners. The findings may help inform future training programs and improve patient care outcomes.

ELIGIBILITY:
Inclusion Criteria:

- Licensed general practitioners actively working primary health care centers, outpatients clinics and general hospitals in Upper Egypt( Assuit, Minya, Sohag, Qena, luxor and Aswan).

Exclusion Criteria:

* Specialists in gastroenterology.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: cross-sectional, observational study.
  Conducted in primary health care centers,
  outpatient clinics, and general hospitals in Up
  Egypt (e.g., Assiut, Sohag, Qena, Minya, Luxo
  Aswan).
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Knowledge | After history and examination by 1 hour.
  Level of knowledge about H. pylori infection among General Practitioners" "Measured using a questionnaire of X items (e.g., 15 multiple-choice questions). The total knowledge score will be calculated as the percentage of correct answers."
Attitudes | After history and examination by 1 hour.
  Attitudes of General Practitioners towards diagnosis and treatment of H. pylori infection" "Measured using an X-point Likert scale (e.g., 5-point) on Y items (e.g., 10 statements). A mean score will be calculated for each participant."
Practices | After history and examination by 1 hour.
  Clinical practices of General Practitioners in managing H. pylori infection" "Measured using questions regarding frequency of testing and types of treatment regimens prescribed. Percentages for each practice will be calculated."
Perceived Barriers | After history and examination by 1 hour.
  Barriers reported by General Practitioners in diagnosing and treating H. pylori infection" "Measured using a checklist or Likert scale containing specific barriers (e.g., lack of resources, time constraints, guideline clarity). Frequencies or scores for each barrier will be calculated."